CLINICAL TRIAL: NCT05253521
Title: The Role of South Asian vs European Origins on Circulating Regenerative Cell Exhaustion
Acronym: ORIGINS-RCE
Status: Completed | Type: Observational
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Collaborators: Unity Health Toronto (Other); Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00059664
Record Dates: First submitted 2022-01-07; First posted 2022-02-23 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Diabetes; Type 1 Diabetes; Type 2 Diabetes; Ischemic Heart Disease; Ischemic Stroke; Cardiovascular Diseases; Peripheral Vascular Diseases
Keywords: Progenitor Cells; Cardiometabolic Risk; Ethnic Origins
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Myocardial Ischemia; Ischemic Stroke; Cardiovascular Diseases; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- South Asian Origin: Individuals who identify as having Anglo-Indian, Bangladeshi, Bengali, Bhutanese, Goan, Gujarati, Indian, Jatt, Kashmiri, Maharashtrian, Malayali, Nepali, Pakistani, Punjabi, Sindhi, Sinhalese, Sri Lankan, Tamil, Telugu, or other South Asian origin
- White Individuals of European Origin: Individuals who identify as having western European, other northern European, southern European, eastern European or other European origin

SUMMARY:
ORIGINS-RCE is an observational, cross-sectional, two-arm study aimed at determining if an individual's ethnic origin influences the number of blood vessel-forming stem cells in the bloodstream. Circulating progenitor cells will be enumerated and the distribution patterns of these cell types will be assessed to determine if these parameters differ between individuals of South Asian origin and European origin. Specifically, this study will evaluate if differential regenerative cell exhaustion (RCE) may account, at least in part, for the differences in cardiovascular risk reported between individuals of South Asian vs European origin.

DETAILED DESCRIPTION:
Individuals of South Asian origins have been reported to be at higher risk of ischemic heart disease than those of European origins. While differential morphometries and culturally related behavioural habits are believed to account in part for the difference, there is growing evidence that cardiometabolic risk factors can accelerate pro-vascular progenitor cell depletion and dysfunction. The cumulative effects that aberrant regenerative cell exhaustion (RCE) have on vessel repair accordingly increases the risk of atherothrombotic events.

ORIGINS-RCE is an observational, cross-sectional, two-arm study that will evaluate the progenitor cell profiles of peripheral blood samples from 120 individuals (60 of South Asian origins, 60 of European origins). The working hypothesis is that individuals of South Asian and European origins have innately different progenitor profiles that can be further altered by behavioural/cultural habits. The resultant differences in RCE capability will affect the balance between pro-inflammatory and vessel repair functions that in turn contribute to the contrasting cardiometabolic risks exhibited between the two study cohorts.

ELIGIBILITY:
1. Adults 40 years of age or older of South Asian origin or white European origin as defined by the following:

   1. South Asian defined as any individual who identifies as Anglo-Indian, Bangladeshi, Bengali, Bhutanese, Goan, Gujarati, Indian, Jatt, Kashmiri, Maharashtrian, Malayali, Nepali, Pakistani, Punjabi, Sindhi, Sinhalese, Sri Lankan, Tamil, Telugu, or other South Asian.
   2. White Europeans or European Origin defined as any individual who identifies as from western European, other northern European, southern European, eastern European or other European origins.
2. Willing and able to provide written informed consent and comply with study requirements.
3. Must meet criteria of one of the two following groups:

   1. Established diabetes (HbA1c ≤10.5%) with no CVD but meets 1 or more of the following criteria:

      * On insulin therapy
      * Cigarette smoker or stopped smoking within 3 months
      * Documented hypertension (as defined by a sitting blood pressure at screening of ≥130/80 mmHg) OR currently on antihypertensive therapy
      * History of treated or untreated dyslipidemia
      * High sensitivity C-reactive protein ≥2.0 mg/L
      * eGFR 30 to 60 mL/min/1.73m^2
      * Documented micro- or macro-albuminuria
   2. Established CVD and meets 1 or more of the following criteria within 10 years prior to screening:

      * Documented coronary artery disease (CAD)
      * Documented cerebrovascular or carotid disease
      * Documented peripheral artery disease (PAD)

Exclusion Criteria:

1. Severe congestive heart failure (as defined by New York Heart Association - class IV)
2. Any life-threatening disease expected to result in death within the next 2 years
3. Any malignancy not considered cured (except basal cell carcinoma of the skin). A subject is considered cured if there has been no evidence of cancer recurrence for the 5 years prior to screening.
4. Known severe liver disease
5. White blood cell count ≥15 x 10^9/L
6. Active infectious disease requiring antibiotic or anti-viral agents
7. Known acquired immunodeficiency syndrome such as HIV
8. On oral steroid therapy (e.g. prednisone or other corticosteroids) or other immunosuppressive agents (e.g. methotrexate)
9. Treated autoimmune disorder (excluding type 1 diabetes)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from primary care and cardiology outpatient clinics in the Greater Toronto Area using paper-based and electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
The change in the frequency / absolute number of circulating ALDHhiSSChi granulocyte precursor cells between individuals of South Asian origins and White individuals of European origin | Baseline

SECONDARY OUTCOMES:
The change in the frequency / absolute number of circulating ALDHhiSSCmid precursor cells with monocytes/macrophage phenotype between individuals of South Asian origins and White individuals of European origin | Baseline
The change in the frequency / absolute number of circulating ALDHhiSSClo cells with primitive provascular progenitor cell phenotype between individuals of South Asian origins and White individuals of European origin | Baseline

OTHER OUTCOMES:
Changes in the concentration of serum oxidative stress markers individuals of South Asian origins and White individuals of European origins | Baseline
Changes in the concentration of serum inflammatory markers individuals of South Asian origins and White individuals of European origins | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, PhD, Principal Investigator — University of Toronto; David A Hess, PhD, Principal Investigator — Western University, Canada
Locations (3):
- Canada (3):
  - Markham HealthPlex Medical Centre, Markham, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Diagnostic Assessment Centre, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sheth T, Nair C, Nargundkar M, Anand S, Yusuf S. Cardiovascular and cancer mortality among Canadians of European, south Asian and Chinese origin from 1979 to 1993: an analysis of 1.2 million deaths. CMAJ. 1999 Jul 27;161(2):132-8. PMID 10439820
- [Background] Misra A, Wasir JS, Pandey RM. An evaluation of candidate definitions of the metabolic syndrome in adult Asian Indians. Diabetes Care. 2005 Feb;28(2):398-403. doi: 10.2337/diacare.28.2.398. PMID 15677799
- [Background] Volgman AS, Palaniappan LS, Aggarwal NT, Gupta M, Khandelwal A, Krishnan AV, Lichtman JH, Mehta LS, Patel HN, Shah KS, Shah SH, Watson KE; American Heart Association Council on Epidemiology and Prevention; Cardiovascular Disease and Stroke in Women and Special Populations Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Stroke Council. Atherosclerotic Cardiovascular Disease in South Asians in the United States: Epidemiology, Risk Factors, and Treatments: A Scientific Statement From the American Heart Association. Circulation. 2018 Jul 3;138(1):e1-e34. doi: 10.1161/CIR.0000000000000580. Epub 2018 May 24. PMID 29794080
- [Background] McKeigue PM, Miller GJ, Marmot MG. Coronary heart disease in south Asians overseas: a review. J Clin Epidemiol. 1989;42(7):597-609. doi: 10.1016/0895-4356(89)90002-4. PMID 2668448
- [Background] Cubbon RM, Murgatroyd SR, Ferguson C, Bowen TS, Rakobowchuk M, Baliga V, Cannon D, Rajwani A, Abbas A, Kahn M, Birch KM, Porter KE, Wheatcroft SB, Rossiter HB, Kearney MT. Human exercise-induced circulating progenitor cell mobilization is nitric oxide-dependent and is blunted in South Asian men. Arterioscler Thromb Vasc Biol. 2010 Apr;30(4):878-84. doi: 10.1161/ATVBAHA.109.201012. Epub 2010 Jan 28. PMID 20110574
- [Background] Putman DM, Liu KY, Broughton HC, Bell GI, Hess DA. Umbilical cord blood-derived aldehyde dehydrogenase-expressing progenitor cells promote recovery from acute ischemic injury. Stem Cells. 2012 Oct;30(10):2248-60. doi: 10.1002/stem.1206. PMID 22899443
- [Background] Hess DA, Wirthlin L, Craft TP, Herrbrich PE, Hohm SA, Lahey R, Eades WC, Creer MH, Nolta JA. Selection based on CD133 and high aldehyde dehydrogenase activity isolates long-term reconstituting human hematopoietic stem cells. Blood. 2006 Mar 1;107(5):2162-9. doi: 10.1182/blood-2005-06-2284. Epub 2005 Nov 3. PMID 16269619
- [Background] Putman DM, Cooper TT, Sherman SE, Seneviratne AK, Hewitt M, Bell GI, Hess DA. Expansion of Umbilical Cord Blood Aldehyde Dehydrogenase Expressing Cells Generates Myeloid Progenitor Cells that Stimulate Limb Revascularization. Stem Cells Transl Med. 2017 Jul;6(7):1607-1619. doi: 10.1002/sctm.16-0472. Epub 2017 Jun 15. PMID 28618138
- [Background] Terenzi DC, Trac JZ, Teoh H, Gerstein HC, Bhatt DL, Al-Omran M, Verma S, Hess DA. Vascular Regenerative Cell Exhaustion in Diabetes: Translational Opportunities to Mitigate Cardiometabolic Risk. Trends Mol Med. 2019 Jul;25(7):640-655. doi: 10.1016/j.molmed.2019.03.006. Epub 2019 Apr 30. PMID 31053416
- [Background] Balber AE. Concise review: aldehyde dehydrogenase bright stem and progenitor cell populations from normal tissues: characteristics, activities, and emerging uses in regenerative medicine. Stem Cells. 2011 Apr;29(4):570-5. doi: 10.1002/stem.613. PMID 21308868
- [Background] Gentry T, Foster S, Winstead L, Deibert E, Fiordalisi M, Balber A. Simultaneous isolation of human BM hematopoietic, endothelial and mesenchymal progenitor cells by flow sorting based on aldehyde dehydrogenase activity: implications for cell therapy. Cytotherapy. 2007;9(3):259-74. doi: 10.1080/14653240701218516. PMID 17464758
- [Background] Shoulars K, Noldner P, Troy JD, Cheatham L, Parrish A, Page K, Gentry T, Balber AE, Kurtzberg J. Development and validation of a rapid, aldehyde dehydrogenase bright-based cord blood potency assay. Blood. 2016 May 12;127(19):2346-54. doi: 10.1182/blood-2015-08-666990. Epub 2016 Mar 11. PMID 26968535
- [Background] Murphy C, Kanaganayagam GS, Jiang B, Chowienczyk PJ, Zbinden R, Saha M, Rahman S, Shah AM, Marber MS, Kearney MT. Vascular dysfunction and reduced circulating endothelial progenitor cells in young healthy UK South Asian men. Arterioscler Thromb Vasc Biol. 2007 Apr;27(4):936-42. doi: 10.1161/01.ATV.0000258788.11372.d0. Epub 2007 Jan 25. PMID 17255539
- [Background] Terenzi DC, Bakbak E, Trac JZ, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Isolation and characterization of circulating pro-vascular progenitor cell subsets from human whole blood samples. STAR Protoc. 2021 Feb 1;2(1):100311. doi: 10.1016/j.xpro.2021.100311. eCollection 2021 Mar 19. PMID 33554145
- [Derived] Park B, Krishnaraj A, Teoh H, Bakbak E, Dennis F, Quan A, Hess DA, Verma S. GLP-1RA therapy increases circulating vascular regenerative cell content in people living with type 2 diabetes. Am J Physiol Heart Circ Physiol. 2024 Aug 1;327(2):H370-H376. doi: 10.1152/ajpheart.00257.2024. Epub 2024 Jun 14. PMID 38874618
- [Derived] Krishnaraj A, Bakbak E, Teoh H, Pan Y, Firoz IN, Pandey AK, Terenzi DC, Verma R, Bari B, Bakbak AI, Kunjummar SP, Yanagawa B, Connelly KA, Mazer CD, Rotstein OD, Quan A, Bhatt DL, McGuire DK, Hess DA, Verma S. Vascular Regenerative Cell Deficiencies in South Asian Adults. J Am Coll Cardiol. 2024 Feb 20;83(7):755-769. doi: 10.1016/j.jacc.2023.12.012. PMID 38355246